CLINICAL TRIAL: NCT04482712
Title: Effects of mTOR Inhibition With Sirolimus (RAPA) in Patients With COVID-19 to Moderate the Progression of Acute Respiratory Distress Syndrome (RAPA-CARDS)
Brief Title: Effects of mTOR Inhibition With Sirolimus (RAPA) in Patients With COVID-19 to Moderate the Progression of ARDS
Acronym: RAPA-CARDS
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was never submitted to IRB or approved, due to feasibility issues
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: The Claude D. Pepper Older Americans Independence Centers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC20200489H
Record Dates: First submitted 2020-07-21; First posted 2020-07-22 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Acute Lung Injury/Acute Respiratory Distress Syndrome (ARDS); Respiratory Failure; Sars-CoV2
Keywords: COVID-19
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome; Respiratory Insufficiency; COVID-19 | interventions — Sirolimus; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a double-blind clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Administration of placebo daily during hospitalization
  Interventions: Drug: Placebo
- Rapamycin (Active Comparator): Administration of rapamycin (sirolimus) 1mg daily during hospitalization
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — Daily administration of a dose of investigational drug for up to 4 weeks while hospitalized
  Other Names: Sirolimus; Rapamune; RAPA
  Arms: Rapamycin
Drug: Placebo — Administration of investigational drug placebo for up to 4 weeks while hospitalized
  Other Names: Placebo Tablet or oral solution
  Arms: Placebo

SUMMARY:
This study assesses the clinical effectiveness of mammalian target of rapamycin (mTOR) inhibition with rapamycin in minimizing or decreasing the severity of acute lung injury/acute respiratory distress syndrome (ALI/ARDS) in participants infected with mild to moderate COVID-19 virus.

DETAILED DESCRIPTION:
This is a single center, double-blind, placebo-controlled, randomized clinical trial in which each participant, after admission to hospital with a diagnosis of mild to moderate COVID-19 infection, will be administered either a dose of rapamycin or the placebo daily. Each subject will receive the assigned treatment until hospital discharge or death. Evaluations will be performed at the beginning of the clinical trial and then daily up to 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Over 60 years of age clinically judged to require hospitalization
2. SARS-CoV2 infection documented by positive RT-PCR nasopharyngeal swab
3. Mild to Moderate clinical status defined as clinical symptoms with or without pneumonia on imaging, with or without fever who are judged to require hospital admission

   1. Elevated ferritin
   2. Lymphopenia
   3. Bilateral opacities on chest x-ray
   4. Low pro-calcitonin
   5. Clinical signs suggestive of symptoms of mild illness with COVID-19 that could include fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms, without shortness of breath or dyspnea or moderate illness with CoVID-19, such as respiratory rate ≥ 20 breaths per minute, saturation of oxygen (SpO2) > 93% on room air at sea level, heart rate ≥ 90 beats per minute.

Exclusion Criteria:

1. Known or suspected allergy to RAPA
2. High pro-calcitonin
3. SARS-CoV2 documented by negative RT-PCR nasopharyngeal swab
4. Treatment with contraindicated concomitant medications: currently receiving immunosuppressants, including steroids, prior to enrollment, or with immunomodulators or immunosuppressant drugs, including but not limited to Inter leukin (IL)-6 inhibitors, Tumor necrosis factor (TNF) inhibitors, anti-IL-1 agents and Janus kinase (JAK) inhibitors within 5 half-lives or 30 days (whichever is longer) prior to randomization.
5. Currently receiving immunosuppressants, including steroids, prior to enrollment
6. Serious underlying disease including but not limited to cardiac, pulmonary, renal, hepatic (bilirubin >1.5x Upper normal limit (ULN) or Aspartate Aminotransferase (AST)>ULN but bilirubin ≤ ULN), endocrine (diabetes) or psychiatric disorders judged to be at risk in participating by the inpatient attending physician or team
7. Suspected or confirmed history of alcohol or substance abuse disorder
8. Having participated in other drug trials in the past month
9. Deemed otherwise unsuitable for the study by researchers
10. Clinically judged to not require hospital admission

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 4 weeks
  The proportion of participants who survive without respiratory failure

SECONDARY OUTCOMES:
Change in Clinical Status assessed by the World Health Organization (WHO) scale | Baseline to 4 weeks
  The WHO ordinal scale is a measure of clinical improvement using a scale score of 0-8, where 0 indicates a better outcome and 8 indicates death:
  Uninfected, no clinical oor virological evidence of infection 0 Ambulatory, no limitation of activities 1 Ambulatory, limitation of activities 2 Hospitalized Mild disease, no oxygen therapy 3 Hospitalized mild disease, oxygen by mask or nasal prongs 4 Hospitalized Severe Disease, non-invasive ventilation 5 Hospitalized severe disease, intubation and mechanical ventilation 6 Hospitalized severe disease, ventilation+organ support 7 Death 8
Change in Clinical Status assessed by the National Institute of Allergy and Infectious Disease (NIAID) scale | Baseline to 4 weeks
  An ordinal scale for clinical improvement scored from 1 to 8, where 1 represents death and 8 represents recovery to discharge from hospital with no limitation on activities:
  Death (1) Hospitalized, on invasive mechanical ventilation of extracorporeal membrane oxygenation (ECMO) (2) Hospitalized, on non-invasive ventilation or high flow oxygen devices (3) Hospitalized, requiring supplemental oxygen (4) Hospitalized, not requiring supplemental oxygen or ongoing medical care (6) Not hospitalized, limitation on activities &/or requiring supplemental home oxygen (7)
  Not hospitalized, no limitation on activities (8)

OTHER OUTCOMES:
All cause mortality | 4 weeks
  Total number of deaths during the study period
Duration of ECMO | Up to 4 weeks
  Number of days on ECMO
Duration of supplemental oxygen | Up to 4 weeks
  Number of days participants are on supplemental oxygen
Length of hospital stay | Up to 4 weeks
  Days of hospitalization
Length of time to SARS-CoV2 negativity | Up to 4 weeks
  Number of days until there is a negative response to the reverse transcriptase-polymerase chain reaction test (RT-PCR)

CONTACTS AND LOCATIONS:
Overall Officials: Dean L Kellogg, MD, PhD, Principal Investigator — University of Texas Health at San Antonio
Locations (2):
- United States (2):
  - University Hospital System, San Antonio, Texas
  - Audie L Murphy Memorial Veterans Hospital, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available at study completion at the time of journal publication.